CLINICAL TRIAL: NCT05871840
Title: Real-World Evidence: Effectiveness and Safety of Repeated Low-Level Red-Light Therapy on Myopia Control Among Children and Adolescents
Brief Title: Effectiveness and Safety of Repeated Low-Level Red-Light Therapy on Myopia Control Among Children and Adolescents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Hospital (Guangming), University of Chinese Academy of Sciences (Other)
Collaborators: the Second of Affiliated Hospital of Wannan Medical College, Wuhu, China (Unknown); First Hospital Affiliated to Baotou Medical College, Baotou, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: LL-KT-2023006-X1
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Treatment duration of RLRL therapy (≥ 6 months and < 12 months)
  Interventions: Other: Repeated Low-Level Red-Light (RLRL) Therapy
- Treatment duration of RLRL therapy (≥12 months and < 24 months)
  Interventions: Other: Repeated Low-Level Red-Light (RLRL) Therapy
- Treatment duration of RLRL therapy (≥24 months and < 36 months)
  Interventions: Other: Repeated Low-Level Red-Light (RLRL) Therapy
- Treatment duration of RLRL therapy (≥36 months)
  Interventions: Other: Repeated Low-Level Red-Light (RLRL) Therapy

INTERVENTIONS:
Other: Repeated Low-Level Red-Light (RLRL) Therapy — This treatment device was made by Eyerising SuzhouXuanjia Optoelectronics Technology, which has been on the market and used widely for amblyopia treatment for the past decade in China. This device is certified as a class IIa device by the China National Medical Products Administration. It consists of semiconductor laser diodes, which deliver low-level red light with a wavelength of 650 ±10 nm at an illuminance level of approximately 1600 lux through the pupil to the fundus. Based on calculations completed by an independent lab, the light power going through a 4-mm pupil is 0.29 mW and is classified as class 1 under the International Electrotechnical Commission 60825-1:2014 standard, which is at a level considered safe for direct ocular exposure that would not create retinal thermal hazard.

SUMMARY:
Myopia has become one of the leading causes of visual impairment globally and brings a heavy burden on the society. Therefore, preventing and controlling the progression of myopia has become an urgent public health issue that needs to be addressed.

The purpose of this study is to provide real-world evidence for identifying the incidence of myopia control (axial length growth rate ≤ 0.1mm/year) after 36-month RLRL therapy, and long-term safety of RLRL therapy in children and adolescents.

DETAILED DESCRIPTION:
The prevalence of myopia in children is increasing worldwide and is viewed as a major public health concern. The current methods for myopia control include medication (e.g., atropine eye drops), optical (e.g., orthokeratology) and environmental interventions (e.g., time outdoors). Nevertheless, these treatments still have limitations. For example, low-concentration atropine may cause systemic side effects and accommodation loss caused by ciliary muscle paralysis. Moreover, the use of orthokeratology in children poses problems such as difficulty wearing, low compliance, and possible complications such as severe corneal infections. Thus, developing the more effective and safe treatment for myopia control in children and adolescents is the future research direction.

Recently, repeated low-level red-light (RLRL) therapy has emerged as a treatment for myopia control in children and adolescents, with promising efficacy and safety. It is suggested that continued RLRL therapy sustained promising efficacy and safety in slowing myopia progression within 2 years. However, relevant information on the effectiveness and safety of RLRL therapy on myopia control over 2 years among children and adolescents remain scarce, which deserves to be further explored.

In this multicenter observational study, the investigators aim to recruit 360 children aged 7-18 years who have currently accepted RLRL therapy at 3 study centers in China. All participants are randomly selected by stratified sampling based on the treatment duration of RLRL therapy (6-12 months, 12-24 months, 24-36 months, 36 months or more). First, the investigators will confirm whether these participants have pre-treatment data (before starting RLRL therapy), including visual acuity, axial length and cycloplegic refraction. Then all the eligible participants who meet the preliminary inclusion criteria, will be invited to come to the corresponding hospitals and further undergo the comprehensive ophthalmic examinations, including visual acuity, measurement of ocular biometric parameters, cycloplegic refraction, slit-lamp examination, color fundus photography, optical coherence tomography (OCT), electroretinography (ERG) and questionnaire surveys.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 7-18 years old
2. Myopia of cycloplegic spherical equivalent refraction (SER) of -1.0D or greater in both of eyes before starting RLRL therapy
3. Participants undergo RLRL therapy currently
4. With complete examination data before starting RLRL therapy, including visual acuity, axial length and cycloplegic spherical equivalence refraction
5. The subject and their guardian voluntarily sign the informed consent form

Exclusion Criteria:

1. Presence of strabismus, binocular vision abnormalities, other ocular abnormalities in either eye
2. Secondary myopia (such as myopia caused by retinopathy of prematurity or other eye diseases in infancy or early childhood) or myopia associated with systemic syndromes (such as Marfan syndrome)
3. Presence of other significant ocular and/or systemic diseases or abnormalities
4. Medical history of previous eye surgery, laser treatment, or intravitreal injection and so on
5. Participants if investigators believe they have contraindications that make them unsuitable for participation.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In this study, the investigators aim to recruit 360 participants aged 7-18 years at 3 study centers from 3 tertiary hospitals in China, stratified by the treatment duration of RLRL therapy including 6 to 12 months (<12 months); 12 to 24 months (< 24 months); 24 to 36 months (< 36 months); and 36 months or more. Thirty participants are recruited at each treatment duration for each study center. Therefore, the minimum number of subjects per study center is 30, and the maximum number of subjects per study center is 120.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of myopia control after 36-month RLRL therapy | 36 months or more
  Validity index: myopia control was defined as axial length growth rate ≤ 0.1mm/year

SECONDARY OUTCOMES:
Incident visual impairment (logMAR visual acuity < 0.8) | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Safety index
Incident structural damage of the retina and choroid | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Safety index
Change of axial length per year after RLRL therapy. | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Validity index
Change of spherical equivalent refraction per year after RLRL therapy | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Validity index
The incidence of myopia control after 6-,12- and 24-month RLRL therapy | 6-12 months, 12-24 months, 24-36 months
  Validity index: myopia control was defined as axial length growth rate ≤ 0.1mm/year
Incident adverse event | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Safety index: adverse events including but not limited to dazzling, short-term glare, flash blindness, and delayed afterimages
Incident severe adverse event | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Safety index: including but not limited to sudden visual loss of >2 lines occurring or a scotoma perceived to develop in the center of the visual field.
Abnormality of the retinal function | 6-12 months, 12-24 months, 24-36 months, 36 months or more
  Safety index: retinal function is evaluated by electroretinogram (ERG)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yu, Principal Investigator — Shenzhen Hospital (Guangming), University of Chinese Academy of Sciences

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as open data after proper anonymization.

REFERENCES:
- [Derived] Chen Y, Wang W, Xiong R, Yu F, Pan S, Dong J, Zhang J, Zhu Z, Ding X, Wang B, Chen Y, Chan HH, Choi KY, Chan SSH, Zheng Y, Shi D, Aung Y, Kishi S, Ohno-Matsui K, He M. Three-year efficacy and safety of repeated low-level red-light therapy for myopia control: a multicentre real-world study. Br J Ophthalmol. 2026 Jan 20:bjo-2025-328687. doi: 10.1136/bjo-2025-328687. Online ahead of print. PMID 41558834